CLINICAL TRIAL: NCT01053650
Title: Placebo Effect of Paracetamol in Healthy Volunteers
Acronym: HOP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0065; 2009-015610-22 (EudraCT Number)
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Open / hidden; Placebo effect
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Paracetamol — Clinical trial conducted in healthy volunteers, prospective, single center, randomized, open / hidden.

SUMMARY:
Paracetamol is one of the most commonly used drugs in the world, indicated for the symptomatic treatment of fever and pain of mild to moderate. More precisely, it is a drug used to relieve pain and reduce fever. The objective of this study is to analyze whether a placebo effect occurs when you take paracetamol for pain, ie if the analgesic effect of paracetamol is partly due to the simple fact of taking a drug.

Moreover, during the study you propose to do a saliva sample, optional, for biological research, pharmacogenetics, to assess how paracetamol is processed and eliminated in your body..

DETAILED DESCRIPTION:
Clinical trial conducted in healthy volunteers, prospective, single center, randomized, open / hidden.

ELIGIBILITY:
Inclusion Criteria:

- Healthy volunteers,

* Aged over 18 years and more than 50 years
* Males,
* Values of vital signs before administration of the test products:
* Systolic between 100-140 mm Hg
* diastolic between 50-90 mm Hg
* cardiac pulse between 45-90 beats per minute
* Free from any treatment in the 7 days preceding inclusion including no use of analgesics or anti-inflammatory)

Exclusion Criteria:

* Contraindications to the administration of paracetamol : Hypersensitivity to paracetamol, History of hepatitis B or C, Severe renal impairment
* Hepatic insufficiency
* Medical history and / or surgical judged by the investigator or his representative as being incompatible with the test, especially subjects with neuropathic pain,
* Pathology evolutionary time of the review of inclusion
* Excessive consumption of alcohol, tobacco (over 10 cigarettes / day), coffee, tea or drinks containing caffeine (equivalent to more than 4 cups per day) or drug abuse,

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The main objective of this protocol is to assess the placebo effect in healthy volunteers by comparing pain thresholds and tolerance between two passages, when taking paracetamol.

SECONDARY OUTCOMES:
The secondary objectives of this study are 1 - explore, through testing Cantab ®, if the administration of paracetamol alter performance on cognitive tests. 2 - to analyze the determination of paracetamol and its metabolites in urine and blood samples,

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, MCU-PH, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France